CLINICAL TRIAL: NCT01547221
Title: Effectiveness of 3% Boric Acid in 70% Alcohol Versus 1% Clotrimazole Solution in Otomycosis Patients: a Randomized Controlled Trial
Brief Title: Effectiveness of 3% Boric Acid in 70% Alcohol Versus 1% Clotrimazole Solution in Otomycosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen Hospital (Other Government)
Responsible Party: Principal Investigator, Ms. Sarisa Romsaithong, Medical physician, senior professional level, Khon Kaen Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KKH24-01-2555
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Otomycosis
Keywords: otomycosis; 3% boric acid; 1% clotrimazole ear drop
MeSH Terms: conditions — Otomycosis | interventions — Clotrimazole; boric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3% boric acid (Active Comparator): control
  Interventions: Drug: 3% Boric acid
- 1% clotrimazole ear drop (Experimental): 3% boric acid is set as control while 1% clotrimazole ear drop is set as intervention.
  Interventions: Drug: clotrimazole

INTERVENTIONS:
Drug: clotrimazole — single application of 1%clotrimazole ear drop
  Other Names: Candid
  Arms: 1% clotrimazole ear drop
Drug: 3% Boric acid — 3% boric acid in 70% alcohol was prepared by phamaceutical department of Khonkaen Hospital
  Arms: 3% boric acid

SUMMARY:
Otomycosis is a superficial fungal infection of the external ear canal. Patients should be treated with cleaning fungal debris combined with topical antifungal agent. There is wide range of topical antifungal agents. However, there is still no consensus of the most effective topical antifungal agents in treatment otomycosis is still lacking.

According to Thai National List of essential medicines for topical antifugal agents are:

* acetic acid (2% in aqueous and 2% in 70% isopropyl alcohol)
* boric acid (3% in isopropyl alcohol)
* gentian violet
* clotrimazole ear drop. But from literature review, there is no comparative study between boric acid and clotrimazole solution before.

Objective is to compare the clinical effectiveness and adverse events of 1% clotrimazole solution versus 3% boric acid in 70% alcohol for the treatment of otomycosis.

DETAILED DESCRIPTION:
The hypothesis has been formulated by H0 and Ha. H0 = 1% clotrimazole solution has clinical effectiveness not different from 3% boric acid in 70% alcohol for the treatment of otomycosis.

Ha = 1% clotrimazole solution has more clinical effectiveness than 3% boric acid in 70% alcohol for the treatment of otomycosis.

Inclusion criteria:

* Symptomatic otomycosis, age more than 7 year.
* Microscopic finding revealed fungus
* KOH smear positive for fungus

Exclusion criteria:

* Pregnancy
* Tympanic membrane perforation and post mastoid surgery
* Co-infection of ear e.g. severe otitis externa,severe myringitis which are needed other medication.
* Previous using topical antibiotic / steroid within 2weeks.
* During usage of systemic antifungal drug
* Allergic to 3% boric acid in 70% alcohol or 1% clotrimazole solution. PICO model: P= otomycosis patient I= 1%clotrimazole ear drop C= 3% boric acid O= result of treatment as cure

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic otomycosis, age more than 7 year.
* Microscopic finding revealed fungus
* KOH smear positive for fungus

Exclusion Criteria:

* Pregnancy
* Tympanic membrane perforation and post mastoid surgery
* Co-infection of ear e.g. severe otitis externa, severe myringitis which are needed other medications
* Previous using topical antibiotic / steroid within 2weeks.
* During usage of systemic antifungal drug
* Allergic to 3% boric acid in70% alcohol or 1% clotrimazole solution.
* Those who can not come to follow up after one week of the treatment

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
result as cure rate of otomycosis | 1 week after treatment
  otolaryngologist's microscopic finding

SECONDARY OUTCOMES:
adverse effect of treatment | Five minutes after apply treatment
  using questionaire to record adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Sarisa Romsaithong, M.D., Principal Investigator — Unaffiliate
Locations (1):
- ENT clinic KhonKaen Hospital, KhonKaen, KhonKaen, Thailand